CLINICAL TRIAL: NCT00299715
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose-Response, Multicenter Study to Evaluate the Efficacy and Safety of Three Fixed Doses of Extended-Release Paliperidone in the Treatment of Subjects With Acute Manic and Mixed Episodes Associated With Bipolar I Disorder
Brief Title: A Study to Evaluate the Efficacy and Safety of Three Fixed Doses of Extended-release Paliperidone in Subjects With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR010834
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Bipolar Disorder; Mood Disorders
Keywords: Affective psychosis; mixed-state; bipolar disorder; manic disorder; manic-depressive; psychosis; mania; manic state; paliperidone; paliperidone ER.
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Affective Disorders, Psychotic; Psychotic Disorders; Mania

INTERVENTIONS:
Drug: Paliperidone extended-release

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of 3 different doses of paliperidone extended release (ER) compared to placebo in patients diagnosed with Bipolar I Disorder who are experiencing an acute manic or mixed episode. This study will also evaluate the effects of paliperidone extended release on global functioning, and the relationship between blood levels and the effectiveness and safety of paliperidone.

DETAILED DESCRIPTION:
Several treatments are available for the treatment of acute manic and mixed episodes associated with bipolar disorder. Some of these treatments although used for many years, are associated with well-known problems such as poor tolerability, significant toxicities, narrow therapeutic ranges, and drug interactions. Often, several drugs must be used in combination to achieve the best clinical effect. More recently, a group of compounds known as atypical antipsychotics, such as risperidone, have been licensed for use in this indication. Based on the pharmacological profile of Paliperidone, it is expected to be effective in the treatment of acute manic and mixed episodes associated with bipolar disorder. Paliperidone extended release has been shown to be effective in schizophrenia and it has an improved drug delivery system with a reduced potential for drug interactions. Study drug tablets are designed to deliver the appropriate amount of drug (3 mg or 6 mg) using a "Push-Pull" delivery system based on a patented oral osmotic pump technology (OROS) that allows the drug to be delivered at a relatively controlled rate for 24 hours. This study will test 3 different doses of paliperidone extended release (3, 6, or 12 mg/day once daily) compared to placebo (inactive substance). There are 3 parts to the study: a screening and washout phase that lasts up to 7 days to determine if patients are eligible for the study and to discontinue all current medications, a double-blind treatment phase that lasts for 3 weeks, and a follow-up phase that lasts about 1 week after the end-of-study visit or early withdrawal from the study. During the double-blind treatment phase, patients are randomly assigned to receive treatment either with placebo or 1 of 3 daily doses of paliperidone extended release. Patients assigned to paliperidone extended release will receive either 3, 6, or 12 mg/day given once daily for a 3-week period. All patients whether receiving paliperidone extended release or placebo will take 2 capsules each time the study drug is given. Patients will be hospitalized for at least the first 7 days of double-blind treatment, and may be discharged on the seventh day and followed as outpatients based on the judgment of the study doctor. End-of-study/early withdrawal procedures will be done after the last dose of study drug has been received and blood samples have been taken, or at early withdrawal from the study. Patients will have a follow-up visit with safety evaluations approximately 1 week later. The study, including the screening and washout phases, will last approximately 35 days or 5 weeks. Effectiveness will be primarily determined by the change in the total Young Mania Rating Scale (YMRS) score from the beginning (baseline) to the end of the double-blind treatment phase of the study. The Young Mania Rating Scale is an 11-item established measure used to evaluate manic symptoms. A secondary measure of effectiveness is the change in the Global Assessment of Functioning Scale (GAF) from baseline to the end of the double-blind treatment phase of the study. Other measures of effectiveness include the time to onset of therapeutic effect, responder rate (defined as 50% or more reduction from baseline in Young Mania Rating Scale score), and changes from baseline to the end of the double-blind treatments phase in all other assessment scales. Additional assessment scales will be used to evaluate the clinical progress of the patient, psychotic and depressive symptoms in bipolar disorder, quality of sleep and daytime drowsiness, health-related function, and rate the severity of the patient's bipolar disorder. Safety will be evaluated by the frequency, severity, and timing of side effects, clinical laboratory tests (including pregnancy tests), 12-lead electrocardiograms (ECGs), vital signs measurements, and physical and neurological examinations. The study hypotheses for the primary and secondary effectiveness measures are 1) that at least 1 dose of paliperidone extended release is better than placebo on the change from baseline in the Young Mania Rating Scale total score at the end of 3 weeks of treatment, and 2) at least 1 dose of paliperidone extended release is better than placebo on the change from baseline in Global Assessment of Functional Scale score at the end of 3 weeks of treatment. The potential effect of the variation in genes related to paliperidone ER may be evaluated separately in patients who consent to DNA (deoxyribonucleic acid) testing. Paliperidone ER, 3, 6, or 12 mg/day or placebo once daily for 3 weeks. To maintain the blind, all patients will take 2 capsules each time study drug is given. Capsules may contain a 3-mg tablet and matching placebo, a 6-mg tablet and matching placebo, two 6-mg tablets, or placebo (inactive) tablets. The doses of study drug will be fixed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM IV) criteria for Bipolar I Disorder, Most Recent Episode Manic or Mixed (with or without psychotic features)
* history of at least 1 previously documented manic or mixed episode requiring medical treatment within 3 years before the screening phase
* total score of at least 20 on the Young Mania Rating Scale at screening and at baseline visit
* if taking mood stabilizers, antipsychotics, or antimanic drugs, must have discontinued that medication at least 3 days before baseline
* women must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent, or agree to practice an effective method of birth control if they are sexually active before entry and throughout the study (effective methods of birth control include prescription hormonal contraceptives, intrauterine devices, double-barrier method, and male partner sterilization)
* able and willing to comply with self-administration of medication, or have consistent help or support available.

Exclusion Criteria:

* Meets Diagnostic and Statistical Manual of Mental Disorders - Fourth Edition criteria for any type of episode associated with Bipolar disorder other than Bipolar I Disorder, Most Recent Episode Manic or Mixed (with or without psychotic features)
* meets DSM-IV criteria for rapid cycling and schizoaffective disorder
* known or suspected borderline or antisocial personality disorder
* in the opinion of the study doctor, is at significant risk for suicidal or violent behavior during the course of the study
* known or suspected history of substance dependence (excluding nicotine and caffeine) within the previous 3 months
* serious or unstable, medical illness (e.g., cardiovascular disease, neurologic, hematologic, renal, immunologic, metabolic, or other systemic illness), or has a history of uncontrolled or insulin-dependent diabetes mellitus
* history of severe, pre-existing gastrointestinal narrowing or inability to swallow study drug with the aid of water
* results at screening or baseline for liver function tests greater than twice the upper limit of the central laboratory reference range
* has active hypo- or hyperthyroidism unless stabilized on appropriate medication for at least 3 months before the screening phase
* history of neuroleptic malignant syndrome
* has a moderate-to-severe degree of tardive dyskinesia at screening
* known or suspected history of hypersensitivity or intolerance to paliperidone or risperidone or suspected history of life-threatening drug allergy or hypersensitivity to any drug
* has received benzodiazepines at doses equal to 4 mg/day of lorazepam or higher for a period of 3 months or longer immediately before the screening phase
* use of clozapine, aripiprazole, or fluoxetine within 1 month before the screening phase
* has received antidepressant therapy, other than fluozetine, within 7 days before the first dose of study drug
* use of antiparkinsonian drugs or beta-blockers (for any indication other than hypertension) within 3 days before the first dose of study drug
* have used cocaine, phencyclidine, amphetamine, methylphenidate, pemoline, an opioid (excluding codeine), hallucinogen, or any other drug that may be associated with manic symptoms as evidenced by a positive urine drug screen
* alcohol intoxication within 3 days before the first dose of study drug
* has had an injection of RISPERDAL CONSTA within 5 weeks before the screening phase, or has received another depot antipsychotic within 1 treatment cycle before the screening phase
* electroconvulsive therapy within 6 months before the first dose of study drug
* women who are pregnant or nursing
* has an anticipated life expectancy of 6 months or less.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The primary effectiveness outcome is the change in the total Young Mania Rating Scale score from baseline to the last assessment during the 3 week double-blind treatment phase.

SECONDARY OUTCOMES:
The secondary effectiveness outcome is the change in Global Assessment of Functional Scale from baseline to endpoint or the last assessment during the double-blind treatment phase.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Berwaerts J, Xu H, Nuamah I, Lim P, Hough D. Evaluation of the efficacy and safety of paliperidone extended-release in the treatment of acute mania: a randomized, double-blind, dose-response study. J Affect Disord. 2012 Jan;136(1-2):e51-e60. doi: 10.1016/j.jad.2010.06.030. Epub 2010 Jul 10. PMID 20624657
- See also: A study to evaluate the efficacy and safety of three fixed doses of extended-release paliperidone in subjects with Bipolar I disorder. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=720&filename=CR010834_CSR.pdf